CLINICAL TRIAL: NCT02325362
Title: Single Center, Double-blind, Randomized, Placebo-controlled, Two-period/Two-treatment Crossover, Proof-of-mechanism Study Investigating the Effect of Miglustat on the Nasal Potential Difference in Adult Patients With Cystic Fibrosis Homozygous for the F508del Mutation
Brief Title: Effect of Miglustat on the Nasal Potential Difference in Patients With Cystic Fibrosis Homozygous for the F508del Mutation
Acronym: MIGLUSTAT-CF
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Actelion (Industry); CRCM (Centres de Ressources et de Compétences de la Mucoviscidose) (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: P120703; 2013-000497-29 (EudraCT Number)
Record Dates: First submitted 2014-12-10; First posted 2014-12-25 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; CFTR; F508del mutation; Miglustat; Total Chloride Secretion; Nasal Potential Difference
MeSH Terms: conditions — Cystic Fibrosis | interventions — miglustat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Miglustat then placebo (Experimental): 10 patients will received Miglustat then the placebo
  Interventions: Drug: Miglustat ; placebo
- Placebo then Miglustat (Experimental): 10 patients will received Placebo then Miglustat
  Interventions: Drug: Placebo ; Miglustat

INTERVENTIONS:
Drug: Miglustat ; placebo — For this 2 x 2 (2 periods /2 treatments) crossover design each patient will receive Miglustat during the first period (2 weeks), following by a wash out period(14 days (up to 4 weeks)), then Placebo during the second period (2 weeks). 30 days follow-up will be carried out after end-of-treatment of the second period.
  Arms: Miglustat then placebo
Drug: Placebo ; Miglustat — For this 2 x 2 (2 periods /2 treatments) crossover design each patient will receive Placebo during the first period (2 weeks), following by wash out period (14 days (up to 4 weeks)), then Miglustat during the second period (2 weeks). 30 days follow-up will be carried out after end of treatment of the second period.
  Arms: Placebo then Miglustat

SUMMARY:
The purpose of this study is to demonstrate that Miglustat restores the function of the cystic fibrosis transmembrane conductance regulator (CFTR) in adult patients with cystic fibrosis homozygous for the F508del mutation.

DETAILED DESCRIPTION:
The aims of this study are:

1. To determine whether Miglustat can restore the function of the CFTR protein in adult patients with cystic fibrosis homozygous for the F508del mutation
2. To evaluate the safety, tolerability and pharmacokinetics of Miglustat in adult patients with cystic fibrosis homozygous for the F508del mutation.
3. To investigate pharmacokinetic-pharmacodynamic of Miglustat in adult patients with cystic fibrosis homozygous for the F508del mutation.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria at screening visit (Visit 1):

* Aged 18 years and older
* Male or female
* Women of childbearing potential must:

  * have a negative serum pregnancy test at Visit 1
  * agree to use from Visit 1 until 3 months after the last study drug intake a reliable method of contraception
* Male patients accepting for the duration of the study and for 3 months thereafter to use a condom
* Homozygous for the F508del mutation as confirmed by genetic testing
* Sweat chloride ≥ 60 mmol/L
* Basal nasal potential difference (NPD) ≤ -30.0 mV (equal to or more electrically negative than -30.0 mV) and total chloride secretion (TCS) ≥ - 5.0 mV for at least one nostril. However, if it is possible to analyze both nostrils, the total chloride secretion (TCS) is to be ≥ - 5.0 mV (equal to or more electrically positive than - 5.0 mV) in both nostrils.
* FEV1 ≥ 25% of predicted
* Able to comply with all protocol requirements
* Signed informed consent prior to any study-mandated procedure

Inclusion criteria at randomization visit (Visit 2):

* Women of child-bearing potential must have a negative urine pregnancy test
* Basal nasal potential difference (NPD) ≤ - 30.0 mV (equal to or more electrically negative than - 30.0 mV) and total chloride secretion (TCS) ≥ - 5.0 mV for at least one nostril. However, if it is possible to analyze both nostrils, the total chloride secretion (TCS) is to be ≥ - 5.0 mV (equal to or more electrically positive than - 5.0 mV) in both nostrils.

Exclusion Criteria:

* Any condition prohibiting the correct measurement of the NPD such as upper respiratory tract infection
* Acute upper or lower respiratory tract infection requiring antibiotic intervention within 2 weeks of screening
* Lung transplant recipient or patient on a lung transplant waiting list
* Any modification in regular treatments (new treatment initiated or discontinued treatment) or modification in dosing within 2 weeks prior to start of Period 1
* Moderate/Severe renal impairment (creatinine clearance < 70 mL/min as per Cockroft and Gault)
* Systemic corticosteroids (> 10 mg/day prednisone or equivalent) within 14 days prior to screening and up to start of study
* Women who are breast-feeding, pregnant, or who plan to become pregnant during the course of the study
* History of significant lactose intolerance
* Presence of clinically significant diarrhoea (> 3 liquid stools per day for > 7 days) without definable cause within one month prior to screening
* Any known factor or disease that might interfere with treatment compliance, study conduct or interpretation of the results such as drug or alcohol dependence or psychiatric disease
* Active or passive smoking
* Hypersensitivity to Miglustat or any excipients
* Planned treatment or treatment with another investigational drug or therapy (e.g., gene therapy) within one month prior to randomization
* Known concomitant life-threatening disease with a life expectancy < 12 months
* Indication against Isuprel® (Isoproterenol) including heart diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-03-17 (Actual); Primary Completion 2017-04-03 (Actual); Study Completion 2017-04-03 (Actual)

PRIMARY OUTCOMES:
Mean TCS in mV | day 1
  TCS (Total Chloride Secretion) is the sum of responses in nasal potential difference (NPD) calculated as the mean of the right and left nostril measurements for each patient
Mean TCS in mV | Day 14
  TCS (Total Chloride Secretion) is the sum of responses in nasal potential difference (NPD) calculated as the mean of the right and left nostril measurements for each patient

SECONDARY OUTCOMES:
TCS difference in mV | day 1
  TCS difference is calculated as the change in measurements of TCS for the right and left nostrils independently for each patient.
TCS difference in mV | Day 14
  TCS difference is calculated as the change in measurements of TCS for the right and left nostrils independently for each patient.
Percentage of patients with a TCS response to treatment ≤ - 5 mV | day 1
  The percentage of patients with a TCS response to treatment defined as a difference in TCS from baseline to end-of-treatment ≤ -5mV
Percentage of patients with a TCS response to treatment ≤ - 5 mV | day 14
  The percentage of patients with a TCS response to treatment defined as a difference in TCS from baseline to end-of-treatment ≤ -5mV
Percentage of patients with a TCS at end-of-treatment ≤ - 5 mV | day 1
  The percentage of patients with a TCS response at end-of-treatment ≤ -5mV
Percentage of patients with a TCS at end-of-treatment ≤ - 5 mV | day 14
  The percentage of patients with a TCS response at end-of-treatment ≤ -5mV
Change of basal NPD in mV | day 1
  Basal NPD at end-of-treatment minus basal NPD at baseline
Change of basal NPD in mV | day 14
  Basal NPD at end-of-treatment minus basal NPD at baseline
Change of the response in NPD after superfusion with amiloride | day 1
  NPD after superfusion with amiloride at end-of-treatment minus NPD after superfusion with amiloride at baseline
Change of the response in NPD after superfusion with amiloride | day 14
  NPD after superfusion with amiloride at end-of-treatment minus NPD after superfusion with amiloride at baseline
Change of the response in NPD after superfusion with a chloride-free buffer in the presence of amiloride | day 1
  NPD after superfusion with a chloride-free buffer in the presence of amiloride at end-of-treatment minus NPD after superfusion with a chloride-free buffer in the presence of amiloride at baseline
Change of the response in NPD after superfusion with a chloride-free buffer in the presence of amiloride | day 14
  NPD after superfusion with a chloride-free buffer in the presence of amiloride at end-of-treatment minus NPD after superfusion with a chloride-free buffer in the presence of amiloride at baseline
Wilschanski's index change | day 1
  Wilschanski's index is defined as (exposant(response to Chloride-free and isoproterenol/response amiloride)): Wilschanski's index at end-of-treatment minus Wilschanski's at baseline
Wilschanski's index change | day 14
  Wilschanski's index is defined as (exposant(response to Chloride-free and isoproterenol/response amiloride)): Wilschanski's index at end-of-treatment minus Wilschanski's at baseline
Sweat chloride concentration in mmol/L | day 1
  Sweat chloride concentration at end-of-treatment minus sweat chloride concentration at baseline
Sweat chloride concentration in mmol/L | day 14
  Sweat chloride concentration at end-of-treatment minus sweat chloride concentration at baseline
FEV1 (in % of predicted) | day 1
  Pulmonary function FEV1: mean Forced expiry volume in 1 second. FEV1 at end-of-treatment minus FEV1 at baseline
FEV1 (in % of predicted) | day 14
  Pulmonary function FEV1: mean Forced expiry volume in 1 second. FEV1 at end-of-treatment minus FEV1 at baseline
Change in electrochemical skin conductance | day 1
  Electrochemical skin conductance at end-of-treatment minus electrochemical skin conductance at baseline
Change in electrochemical skin conductance | day 14
  Electrochemical skin conductance at end-of-treatment minus electrochemical skin conductance at baseline
Number of cells expressing CFTR at the cell membrane (in %percentage) | day 14
  Percentage of nasal cells expressing CFTR at the cell membrane as assessed by immunochemistry and confocal microscopy

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle FAJAC, MD, PhD., Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Assistance publique-Hôpitaux de Paris, Hôpital Cochin, Paris, France

IPD SHARING:
Plan to Share IPD: No